CLINICAL TRIAL: NCT06237946
Title: A Retrospective, Open-label, Biomarker Study for Early-stage Ovarian Clear Cell Carcinoma (OCCC) Patients at Risk of Recurrence
Brief Title: Early-stage Ovarian Clear Cell Carcinoma (OCCC) Patients at Risk of Recurrence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Tokyo University (Other); Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 202310152RIND
Record Dates: First submitted 2024-01-11; First posted 2024-02-02 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: FIGO Stage IC2 to II Ovarian Clear Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine the risk of recurrence in early-stage OCCC (Ovarian Clear Cell Carcinoma) patients who received postoperative adjuvant treatment.

Participants were received platinum-based adjuvant therapy following debulking surgery will be included for the study.

DETAILED DESCRIPTION:
This is a retrospective, global multicenter, single-arm, study for early-stage OCCC (Ovarian Clear Cell Carcinoma) patients at risk of recurrence following the first-line treatment. This study is planned to enroll 272 patients eligible for participation from two study sites in Taiwan, one in Korea, and one in Japan. The study will use archival Formalin-Fixed Paraffin-Embedded (FFPE) samples from patients who have received adjuvant therapy following debulking surgery. The study is designed to identify OCCC patients at risk for relapse and apply clinical stratification by IHC staining of 3 selected markers (CD45, CD8, tryptase) to prepare as clinical assays.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥20 years old.
* Participant with histologically confirmed OCCC of stage IC2, IC3, IIA and IIB by International Federation of Gynecology and Obstetrics (FIGO) 2014 system.
* Participant has received platinum-based regimens for 3 to 6 cycles combined with paclitaxel, gemcitabine, cyclophosphamide, or bevacizumab adjuvant therapy following debulking surgery.
* Formalin-fixed paraffin-embedded (FFPE) tissue samples available.

Exclusion Criteria:

* Absence of histological confirmation of the diagnosis.
* Unusable sample or biologically deteriorated.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 272 women with a diagnosis of FIGO stage IC2, IC3, IIA and IIB of OCCC, diagnosed between 2011 and 2021. Patients were received platinum-based adjuvant therapy following debulking surgery will be included for the study. Adjuvant therapy was given according to the NCCN guideline and Institutional Tumor Board.
Sampling Method: Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of recurrence | up to 24 months
  The clinical recurrence will be defined as disease progression. Analysis of the eligible histologically confirmed OCCC archival samples from Taiwan, Japan, and Korea that underwent immune-related gene expression will be provided.

SECONDARY OUTCOMES:
2-year PFS | up to 24 months
  PFS will be defined as the interval from the surgery date to clinically defined recurrence, disease progression or the last follow-up. PFS will be analyzed using the Kaplan-Meier method, and survival curves will be provided.
5-year OS | up to 60 months
  OS will be calculated from the surgery date to the date of death or the last follow-up. OS will be analyzed using the Kaplan-Meier method, and survival curves will be provided.
Outcomes for adjuvant treatment with paclitaxel-based chemotherapy | up to 60 months
  Hazard ratio (HR) will be evaluated. These data will be analyzed using the Cox proportional hazards model and the Multivariable Cox proportional hazards model.

IPD SHARING:
Plan to Share IPD: No